CLINICAL TRIAL: NCT03950349
Title: FUSION EVALUATION AFTER ANTERIOR CERVICAL DISCECTOMY AND FUSION WITH STAND ALONE LOCKING CAGE WITH BLADE HRCC®
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: PO18157
Record Dates: First submitted 2019-05-13; First posted 2019-05-15 (Actual); Last update posted 2019-05-15 (Actual); Status verified 2019-04

CONDITIONS: Cervical Radiculopathy; Cervical Spinal Fusion; Cervical Myelopathy
Keywords: Radiculopathy; myelopathy; anterior cervical fusion; stand-alone cage; pseudoarthrosis; stabilization; HRCC
MeSH Terms: conditions — Radiculopathy; Klippel-Feil Syndrome; Spinal Cord Diseases; Pseudarthrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- "Anterior cervical discectomy" group

SUMMARY:
Cervical degenerative disease is an almost universal concomitant of human aging. Over half of the middle aged population has cervical spondylosis. This condition is often asymptomatic, but in 10% to 15% of the cases, it is associated with, or progresses to, neural compression. Cervical spondylotic radiculopathy is a condition due to a root nerve compression while cervical spondylotic myelopathy is a condition due to a medullar cord compression. Root nerve or medullar cord can be compressed either by a soft disc extrusion or by arthrosis due to a degenerative disc. Anterior cervical discectomy and fusion is the standard surgical treatment of the cervical radiculopathy or cervical myelopathy when non-surgical treatment failed. The aim of this surgery is to provide a neurologic decompression associated to spine stabilization. Decompression is achieved by removal the disc and soft disc extrusion if present. Stabilization is supported by implantation of material in the interbody space like bone or cage with bone substitute. This cage provides a bone fusion matrix and an intervertebral height and stability support at the same time. To enforce the stabilization, a plate can be screwed on the anterior cervical vertebral wall. The HRCC® cage is a stand-alone cage with two rotary blades which penetrate into vertebral bone so there is no need to implant plate. One of the reasons why treatment can fail is the pseudarthrosis that is fusion failure. It mays occur as an increase of axial pain or radicular pain. The aim of this study is to demonstrate similar results on bone fusion in the surgical treatment of cervical radiculopathy or myelopathy with HRCC cage used in anterior cervical discectomy and fusion compared with other technics based on a prospective cohort study and a literature review. As secondary outcomes we will search to correlate pseudarthrosis and quality of life impact, to identify complications and to describe the sagittal balance evolution of the cervical spine. To this end, in the context of standard practices, patients who consult the neurosurgical team of the REIMS University Hospital Center with a diagnosis of a cervical radiculopathy or myelopathy with non-surgical treatment failure needing a one level anterior cervical discectomy and fusion will be proposed to be included during this pre-operative consultation. There will be pre-operative collected data about demographic data, pseudarthrosis risk factors, pre-operative symptomatology, quality of life data and pre-operative imagery data. Per-operative and hospitalization data are collected as well with surgery duration, blood lost, surgical technic, pain measurement and hospitalization duration. Next, follow-up starts with consultations at 6 weeks, 6 months and 12 months and pain, quality of life and classic X-Ray data are collected to be compared with pre-operative data. And Imagery data are collected in order to identify presence or absence of pseudarthrosis with dynamic X-Ray and CT-scan at 6 months and 12 months. A statistical analysis of the data is next performed to found significant results.

DETAILED DESCRIPTION:
Introduction:

Cervical degenerative disease is an almost universal concomitant of human aging. Over half of the middle aged population has radiological or pathological evidence of cervical spondylosis. This condition is often asymptomatic, but in 10% to 15% of the cases, it is associated with, or progresses to, neural compression. Cervical spondylotic radiculopathy is a condition due to a root nerve compression while cervical spondylotic myelopathy is a condition due to a medullar cord compression. Root nerve or medullar cord can be compressed either by a soft disc extrusion or by osteophyte due to a degenerative disc. Anterior cervical discectomy and fusion is the gold standard treatment of those conditions when non-surgical treatment failed. The aim of this surgery is to provide a neurologic decompression associated to an intervertebral segmental stabilization. Decompression is achieved by discectomy and stabilization by cervical interbody bone fusion. This bone fusion is supported by implantation of material in the interbody space like bone or Poly-Ether-Ether-Keton cage with bone substitute. This cage provides a bone fusion matrix and an intervertebral height and stability support at the same time. To enforce the stabilization, a plate can be screwed on the anterior cervical vertebral wall. The HRCC® cage is a stand-alone cage with no need to implant plate. One risk of this technic is the secondary migration of the cage. That's why this cage is maintained with two rotary blades which penetrate into vertebral plates. It allows easier surgical procedure, with a lower duration of surgery. But one of the reasons of treatment failure is pseudarthrosis. It is defined as the absence of bone bridging the fusion area without any lucencies. It mays occur as an increase of axial pain or radicular pain. The aim of this study is to demonstrate similar results on bone fusion in the surgical treatment of cervical radiculopathy or myelopathy with HRCC cage used in anterior cervical discectomy and fusion compared with other technics based on a prospective cohort study and a literature review.

Materiel and Method In the context of standard practices, patients are included in the study when they consult the neurosurgical team of the REIMS University Hospital Center with diagnosis of one level cervical discopathy causing cervical radiculopathy or myelopathy with non-surgical treatment failure needing a one level anterior cervical discectomy and fusion. Patients are proposed to be included during this pre-operative consultation and they are informed about the protocol and the data collected. If they accept it and sign the non-opposition form, they are included in the study.

The collected data at the pre-operative consult are classic demographic data with age and sex, clinic data with weight, height and BMI, pseudarthrosis risk factors with diabete, tobacco addiction, chronic use of corticosteroid and osteoporosis with confirmed diagnosis, pre-operative symptomatology with presence of cervical radiculopathy with or without deficit, cervical myelopathy with or without pyramidal syndrome at the inferior limb and measurement of neck and radicular arm pain using a numeric scale, quality of life data with the Neck Disability Index (NDI) and the 12-Item Short Form Survey (SF-12), pre-operative imagery data with cervical IRM and the discopathy level, with cervical X-Ray in the profile incidence and measurement of cervical lordosis, measurement of regional lordosis, height. Per-operative collected data are duration of surgery, bleeding, used bone graft either allograft or autograft and final arthrodesis level. Immediate post-operative data are collected the last day of hospitalization with measurement of neck and arm pain using a numeric scale, complications with dysphagia, dysphonia, cervical compressive hematoma with urgent surgical revision, motor neurological deficit with rating if present, surgical revision, duration of the hospitalization in days, post-operative imagery data with cervical lordosis, regional lordosis, height as previously describe, and cage migration. There is a 12 months follow-up with consultations at 6 weeks, 6 months and 12 months. Collected data are for all measurement of neck and radicular arm pain using a numeric scale for the neck and for the arm, persistence of complications with dysphagia, dysphonia, and motor neurological deficit with rating if present, imagery data with cervical lordosis, regional lordosis, height as previously describe, and cage migration. At 6 months and 12 months we add quality of life data with the NDI and the SF-12, dynamic cervical X-Ray data with the measurement of the spinous process shift and CT-scan data. The diagnosis of pseudarthrosis is established on this multimodal imagery. As secondary outcomes, we will search to correlate pseudarthrosis and quality of life impact, to identify complications and to describe the sagittal balance evolution of the cervical spine.

Then, when all the data will be collected, statistical analyses will be performed with description of the cohort and descriptive statistics of all the demographic, radiographic and clinical parameters detailed above for the whole cohort: Mean (±SD) for the continuous variables and Median (±IQR) for the categorical variables. A comparison between pseudarthrosis group and fused group will be performed with univariate analysis (Student test, Wilcoxon test, Chi2 or Exact Fisher test) then a multivariate analysis will be performed with a logistic regression.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of one level cervical discopathy causing cervical radiculopathy or myelopathy with non-surgical treatment failure needing a one level anterior cervical discectomy and fusion
* Age > 18 years old
* Agree to take part at this study

Exclusion Criteria:

* More than one intervertebral level needs to be fused
* Antecedent of spine cervical fracture
* Active cervical malignancy
* Antecedent of cervical spine surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who consult the neurosurgical team of the REIMS University Hospital Center with diagnosis of one level cervical discopathy causing cervical radiculopathy or myelopathy with non-surgical treatment failure needing a one level anterior cervical discectomy and fusion.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-07-01 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
Pseudarthrosis | 6 months
  Pseudarthrosis diagnosis is comfirmed if :
  * CT-scan documents an absence of bone bridging in the extra-graft area
  * measurement of the spinous process shift which is the difference between the inter-spinous process distance on the flexion image and the inter-spinous process distance on the extension image. It is positive when it is more than 1mm at the arthrodesis level associated with a more than 4mm spine process shift at adjacent superior and inferior levels on dynamic cervical X-Ray.
Pseudarthrosis | 12 months
  Pseudarthrosis diagnosis is comfirmed if :
  * CT-scan documents an absence of bone bridging in the extra-graft area
  * measurement of the spinous process shift which is the difference between the inter-spinous process distance on the flexion image and the inter-spinous process distance on the extension image. It is positive when it is more than 1mm at the arthrodesis level associated with a more than 4mm spine process shift at adjacent superior and inferior levels on dynamic cervical X-Ray.

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France